CLINICAL TRIAL: NCT01962870
Title: Randomized Placebo-controlled Trial of Vasopressin Treatment for Social Deficits in Children With Autism
Brief Title: The Role of Vasopressin in the Social Deficits of Autism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Antonio Hardan, MD, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB-26034; R21MH100387-01 (NIH)
Record Dates: First submitted 2013-10-08; First posted 2013-10-14 (Estimated); Results first posted 2019-05-24 (Actual); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: Autism Spectrum Disorders
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Vasopressins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo Nasal Spray
  Interventions: Drug: Placebo
- Vasopressin (Active Comparator): Vasopressin Nasal Spray
  Interventions: Drug: Vasopressin

INTERVENTIONS:
Drug: Vasopressin — Participants aged 6 to 9.5 years of age will receive the maximum dose of 24 IU (12 IU twice daily). Participants aged 9.6 to 12 years of age will receive the maximum dose of 32 IU (16 IU twice daily).
  Arms: Vasopressin
Drug: Placebo
  Arms: Placebo

SUMMARY:
Researchers at the Stanford University School of Medicine are seeking participants for a study examining the effectiveness of vasopressin, a neuropeptide, in treating children with autism spectrum disorder. Difficulty with social interactions is characteristic of people with autism, who often have problems interpreting facial expressions or maintaining eye contact while talking with someone. There are currently no effective medicines available to treat social problems in individuals with autism. Neuropeptides, such as vasopressin and oxytocin, are molecules used by neurons in the brain to communicate with one another. Vasopressin is closely related to oxytocin, which is currently being tested as a treatment for autism, and has been shown to enhance social functioning in animals. Animal studies have shown that when the proper functioning of vasopressin is experimentally altered, animals develop a variety of social deficits, including impaired memory for peers and a reduced interest in social interaction. Researchers found that when vasopressin was administered to mice with a genetically induced form of autism, their social functioning improved. Vasopressin is already approved by the Food and Drug Administration for use in humans, and has proved to be a successful treatment for some common pediatric conditions, including bedwetting. Similar to oxytocin, it also has been shown to improve social cognition and memory in people who do not have autism. The researchers will test the effects of vasopressin on social impairments in 50 boys and girls with autism, ages 6 to 12 years old. The study will last four weeks for each participant. Participants will receive either vasopressin or a placebo nasal spray. At the end of this phase of the study, those who received the placebo will have the option of participating in a four-week trial during which they will be given vasopressin. Stanford is the only site for the study. Participants do not need to live locally but will need to come to the Stanford University Department of Psychiatry and Behavioral Sciences for study visits.

ELIGIBILITY:
Inclusion Criteria:

* medically healthy outpatients between 6 and 12 years of age (cut off: 12 years and 11 months)
* Intelligence Quotient (IQ) equal to or greater than 50 (Stanford-Binet)
* Social Responsiveness Scale (SRS) Total Score equal to or greater than 70
* ability to complete laboratory and cognitive testing
* diagnosis of Autism Spectrum Disorder (ASD) based on expert clinical opinion and confirmed on the Autism Diagnostic Interview-Revised (ADI-R), Autism Diagnostic Observation Schedule (ADOS)
* Clinical Global Impression (CGI) severity rating of 4 or higher
* care provider who can reliably bring participant to clinic visits, provide trustworthy ratings, and interact with the participant on a regular basis
* stable medications for at least 4 weeks
* no planned changes in psychosocial interventions during the trial
* no concurrent participation in any other clinical research trials
* willingness to provide blood samples and electrocardiogram

Exclusion Criteria:

* diagnosis of schizophrenia, schizoaffective disorder, bipolar disorder, or psychotic disorder
* regular nasal obstruction or nosebleeds
* active and unstable medical problems (e.g., migraine; asthma; seizure disorder; anaphylaxis; epilepsy; diabetes; serious liver, renal, or cardiac pathology)
* clinically significant abnormal vital signs or ECG reading
* evidence of a genetic mutation know to cause ASD (e.g., Fragile X Syndrome) or metabolic disorder
* significant hearing or vision impairments
* drinks large volumes of water (e.g., habitual or psychogenic polydipsia)
* pregnant or sexually active females not using a reliable method of contraception (urine pregnancy test will be conducted)
* history of hypersensitivity to vasopressin, its analogs (e.g., Desmopressin), or compounding preservatives (e.g., chlorobutanol)
* current use of any medications known to interact with vasopressin including: 1) carbamazepine (i.e., Tegretol); chlorpropamide; clofibrate; urea; fludrocortisone; tricyclic antidepressants (all of which may potentiate the antidiuretic effect of vasopressin when used concurrently); 2) demeclocycline; norepinephrine; lithium; heparin; alcohol (all of which may decrease the antidiuretic effect of vasopressin when used concurrently); 3) ganglionic blocking agents including benzohexonium, chlorisondamine, pentamine (all of which may produce a marked increase in sensitivity to the pressor effects of vasopressin)
* prior or current use of vasopressin
* abnormal chemistry result

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2017-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Y Hardan, MD, Principal Investigator — Stanford University; Karen J Parker, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine; Psychiatry and Behavioral Sciences, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Iffland M, Livingstone N, Jorgensen M, Hazell P, Gillies D. Pharmacological intervention for irritability, aggression, and self-injury in autism spectrum disorder (ASD). Cochrane Database Syst Rev. 2023 Oct 9;10(10):CD011769. doi: 10.1002/14651858.CD011769.pub2. PMID 37811711

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in the Autism and Developmental Disorders Clinic in the Division of Child and Adolescent Psychiatry at Stanford University. Recruitment began in December 2013 and ended in May 2017.
Pre-assignment Details: 68 participants signed the consent form and enrolled in the study. Of those 68 participants, 27 participants did not meet the eligibility criteria for the study and 11 participants declined to participate prior to randomization. 30 participants were randomized.
Groups:
- Placebo: Placebo Nasal Spray
  Placebo
Period: Overall Study
Arm/Group | Placebo | Vasopressin
Started | 13 | 17
Completed | 13 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants who were randomized in the trial.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Vasopressin | Total
Number analyzed (Participants) | 13 | 17 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 13 | 17 | 30
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 11 | 14 | 25
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 11 | 8 | 19
  Other | 2 | 9 | 11
Region of Enrollment [Number; unit: participants]
  United States | 13 | 17 | 30

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Parent Rated Social Responsiveness Scale, 2nd Edition (SRS-2) T-Score After Treatment.
Description: Social Responsiveness Scale, 2nd Edition (SRS) scores measure social abilities with lower scores meaning better social abilities. (T-Score Range: 37- above 90 )
Time Frame: Baseline; Week 4
Population: Participants who completed the protocol are included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Vasopressin
Number analyzed (Participants) | 13 | 17
units on a scale | 10.8 (2.11) | 17.6 (1.37)

2. Secondary Outcome: Change From Baseline in Clinical Global Impression (CGI) Severity, Social and Communication Scores During Treatment.
Description: Higher Scores on the CGI severity scale mean more greater social and communication deficits (Range 1-7)
Time Frame: Baseline; Week 4
Population: Participants with available data are included.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Vasopressin
Number analyzed (Participants) | 13 | 17
units on a scale | 0.712 (0.202) | 0.873 (0.126)

3. Secondary Outcome: Change From Baseline in Reading the Mind in the Eyes Test, Child Version (RMET-child) Scores During Treatment.
Description: Higher scores mean better ability to read emotions and lower scores mean worse ability to read emotions. Range 0-28.
Time Frame: Baseline; Week 4
Population: Participants with available data are included in the analysis.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Vasopressin
Number analyzed (Participants) | 13 | 17
units on a scale | -1.28 (1.24) | 4.04 (1.63)

4. Secondary Outcome: Change From Baseline in Laboratory Based Facial Emotion Recognition Abilities During Treatment.
Description: Higher scores mean better facial emotion recognition abilities. Lower scores mean worse facial emotion recognition abilities (Range: 0-42).
Time Frame: Baseline; Week 4
Population: Participants with available data are included in the analysis.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Vasopressin
Number analyzed (Participants) | 13 | 17
units on a scale | -7.19 (1.81) | 3.10 (2.42)

5. Secondary Outcome: Change From Baseline in Parent Rated Repetitive Behavior Scale Revised (RBS-R) Scores During Treatment.
Description: Higher scores on the Repetitive Behavior Scale- Revised mean higher levels of repetitive and restricted behaviors. (Raw Score Total Range: 0 - 129)
Time Frame: Baseline; Week 4
Population: Participants with available data were analyzed.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Vasopressin
Number analyzed (Participants) | 13 | 17
units on a scale | 21.3 (3.18) | 17.2 (1.83)

6. Secondary Outcome: Change From Baseline in Parent Rated Spence Children's Anxiety Scale (SCAS) During Treatment.
Description: Scale measuring severity of anxiety symptoms. Higher scores mean higher levels of anxiety, lower scores mean lower levels of anxiety. (Raw Score Range: 0 - 114)
Time Frame: Baseline; Week 4
Population: Participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Vasopressin
Number analyzed (Participants) | 13 | 17
units on a scale | 9.14 (2.68) | 17.9 (1.66)

7. Secondary Outcome: Number of Participants With Side Effects Assessed Using Parent Rated Dosage Record Treatment Emergent Symptom Scale (DOTES) Scores During Treatment
Description: Dosage Record Treatment Emergent Symptom Scale (DOTES) side effects reported by parents during 4-weeks of treatment. Participant Counts are used.
Time Frame: Baseline through Week 4
Population: Participants who completed the protocol are included in the analysis.
Measure: Number; unit: participants
Arm/Group | Placebo | Vasopressin
Number analyzed (Participants) | 13 | 17
participants
  Fever | 1 | 2
  Cough | 0 | 1
  Body Ache | 0 | 1
  Excitement/Agitation | 1 | 0
  Insomnia | 1 | 4
  Increased Motor Activity | 0 | 4
  Depressive Affect | 1 | 2
  Headache | 0 | 2
  Drowsiness | 3 | 1
  Decreased Motor Activity | 2 | 1
  Aggression | 1 | 1
  Akathisia | 0 | 1
  Head Banging | 0 | 1
  Dizziness | 1 | 0
  Lethargy/Tiredness | 1 | 0
  Nasal Congestion | 4 | 3
  Dry Mouth | 3 | 1
  Blurred Vision | 1 | 1
  Ear Infection | 1 | 0
  Runny Nose | 1 | 0
  Sore Throat | 1 | 0
  Cold Sore | 1 | 0
  Decreased Appetite | 5 | 4
  Nausea/Vomiting | 2 | 2
  Constipation | 0 | 1
  Diarrhea | 1 | 0
  Increased Urination | 1 | 1
  Bed Wetting | 0 | 1
  Skin Rash | 1 | 1
  Bug Bite | 0 | 1
  Skin Burn | 1 | 0

8. Secondary Outcome: Change From Baseline on the Overt Aggression Scale (OAS) During Treatment.
Description: Count of participants reporting an increase of aggression during treatment compared to baseline (pretreatment).
Time Frame: Baseline through Week 4
Population: Participants with available data are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Vasopressin
Number analyzed (Participants) | 13 | 17
Participants | 1 | 1

9. Secondary Outcome: Change From Baseline in Heart Rate After Treatment.
Description: Sitting heart rate (beats per minute).
Time Frame: Baseline; Week 4
Population: Participants who completed the protocol are included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Beats per minute
Arm/Group | Placebo | Vasopressin
Number analyzed (Participants) | 13 | 17
Beats per minute | 7.5 (4.43) | 1.9 (3.87)

10. Secondary Outcome: Change From Baseline in Parent Rated Aberrant Behavior Checklist (ABC) Scores During Treatment.
Description: Higher scores indicate more symptoms, lower scores indicate fewer symptoms. Irritability scores can range from 0-45. Lethargy scores can range from 0-48. Stereotypy scores can range from 0-21. Hyperactivity scores can range from 0-48. Inappropriate speech scores can from 0-12.
Time Frame: Baseline; Week 4
Population: Participants with available data were included in analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Vasopressin
Number analyzed (Participants) | 13 | 17
units on a scale
  Irritability Baseline | 14.00 (10.23) | 8.29 (7.40)
  Irritability Week 4 | 8.38 (7.23) | 6.24 (7.05)
  Lethargy Baseline | 14.77 (10.69) | 10.76 (6.32)
  Lethargy Week 4 | 12.77 (9.81) | 7.41 (6.88)
  Stereotypy Baseline | 5.08 (5.36) | 5.18 (3.88)
  Stereotypy Week 4 | 4.54 (4.91) | 3.53 (3.59)
  Hyperactivity Baseline | 21.38 (9.17) | 16.00 (11.69)
  Hyperactivity Week 4 | 14.54 (7.34) | 12.29 (9.06)
  Inappropriate Speech Baseline | 4.62 (3.74) | 3.94 (2.86)
  Inappropriate Speech Week 4 | 3.69 (3.52) | 3.41 (3.08)

11. Secondary Outcome: Change From Baseline in Parent Rated Pediatric Quality of Life (PedQL) Inventory Scores During Treatment.
Description: Higher scores mean better quality of life and lower scores mean worse quality of life (Range: Minimum=0; Maximum=100).
Time Frame: Baseline; Week 4
Population: Participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Vasopressin
Number analyzed (Participants) | 13 | 17
units on a scale
  Baseline | 57.14 (16.67) | 64.53 (13.86)
  Week 4 | 65.96 (14.93) | 74.52 (15.38)

12. Secondary Outcome: Change From Baseline in Parent Rated Vineland Adaptive Behavior Scales Second Edition (VABS-II) - Social and Communication Subscales During Treatment.
Description: Higher Social Standard Score means better social skills, lower Social Standard Score means worse social skills. Higher Communication Standard Score means better communication skills, lower Communication Standard Score means worse communication skills. Standard Scores can range from 20 to 160.
Time Frame: Baseline; Week 4
Population: Not all participants were able to fully complete the measure so not all of the numbers analyzed are the same.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Vasopressin
Number analyzed (Participants) | 13 | 17
units on a scale
  Baseline Social Standard Score: number analyzed (Participants) | 9 | 12
  Baseline Social Standard Score | 61.33 (13.93) | 71.08 (14.38)
  Week 4 Social Standard Score: number analyzed (Participants) | 8 | 15
  Week 4 Social Standard Score | 62.25 (7.78) | 79.67 (16.83)
  Baseline Communication Standard Score: number analyzed (Participants) | 9 | 13
  Baseline Communication Standard Score | 75.67 (13.57) | 74.77 (8.60)
  Week 4 Communication Standard Score: number analyzed (Participants) | 10 | 17
  Week 4 Communication Standard Score | 77.40 (10.55) | 81.12 (14.26)

13. Secondary Outcome: Change From Baseline in Clinical Chemistry Labs (NA+, K+, Cl-) During Treatment.
Description: Clinical chemistry labs(sodium, potassium, chloride)
Time Frame: Baseline; Week 4
Population: Participants with available data are included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Placebo | Vasopressin
Number analyzed (Participants) | 13 | 17
mmol/L
  Change From Baseline in Sodium | 0.15 (0.72) | 0.24 (0.63)
  Change from Baseline in Potassium | 0.06 (0.13) | 0.15 (0.11)
  Change from Baseline on Chloride | -0.31 (0.64) | 1.0 (0.56)

14. Secondary Outcome: Change From Baseline in Laboratory Based Eye-gaze to Social Cues During Treatment.
Time Frame: Baseline; Week 4
Population: Data were not not collected for this outcome.
Arm/Group | Placebo | Vasopressin
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Change From Baseline in Laboratory Based Social Mimicry Abilities During Treatment.
Time Frame: Baseline; Week 4
Population: Data were not not collected for this outcome.
Arm/Group | Placebo | Vasopressin
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Change From Baseline in Blood Pressure After Treatment
Description: Sitting Systolic and Diastolic blood pressure.
Time Frame: Baseline; Week 4
Population: Participants with available data are included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: mmHG
Arm/Group | Placebo | Vasopressin
Number analyzed (Participants) | 13 | 17
mmHG
  Change from Baseline in Systolic Blood Pressure | -1.1 (2.89) | 5.5 (2.53)
  Change from Baseline in Diastolic Blood Pressure | -1.8 (2.39) | 3.2 (2.09)

17. Secondary Outcome: Change From Baseline in Body Weight After Treatment.
Time Frame: Baseline; Week 4
Population: Participants with available data are included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: kilograms
Arm/Group | Placebo | Vasopressin
Number analyzed (Participants) | 13 | 17
kilograms | 0.2 (0.34) | 0.3 (0.30)

18. Secondary Outcome: Change From Baseline in Body Temperature After Treatment
Time Frame: Baseline; Week 4
Population: Participants with available data are included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Degrees (Farenheit)
Arm/Group | Placebo | Vasopressin
Number analyzed (Participants) | 13 | 17
Degrees (Farenheit) | -0.2 (0.19) | 0.2 (0.17)

19. Secondary Outcome: Change From Baseline in the Awareness of Social Inference Test Revised (TASIT-R) Scores During Treatment.
Time Frame: Baseline, Week 4
Population: Data were not not collected for this outcome.
Arm/Group | Placebo | Vasopressin
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Change From Baseline in a Developmental Neuropsychological Assessment, Second Edition. (NEPSY-II) Affect Recognition Scores During Treatment.
Description: Higher Affect Recognition scores mean better affect recognition abilities, lower Affect Recognition scores mean worse affect recognition abilities.
  Scores can range from 1 to 19.
Time Frame: Baseline; Week 4
Population: Participants with available data were included.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Vasopressin
Number analyzed (Participants) | 13 | 17
units on a scale | -2.58 (1.9) | 0.094 (2.20)

21. Secondary Outcome: Change From Baseline in Plasma Vasopressin Levels During Treatment.
Description: There are no clinical laboratory tests that establish a normative range for vasopressin. Measurements prior to treatment were intended to evaluate vasopressin level as a predictor of response. Plasma vasopressin levels post treatment were not quantified. Baseline vasopressin levels are included in the outcome data below.
Time Frame: Baseline
Population: Participants with available data were included in the analysis.
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Placebo | Vasopressin
Number analyzed (Participants) | 13 | 17
pg/ml | 1.28 (0.29) | 1.32 (0.25)

ADVERSE EVENTS:
Time Frame: 4 weeks
Description: Dosage Record Treatment Emergent Symptom Scale (DOTES) and Overt Aggression Scale (OAS) were used to assess side effects.
Arm/Group | Placebo | Vasopressin
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/17
Other Adverse Events (participants affected / at risk) | 12/13 | 13/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=13) | Vasopressin (N=17)
Fever (General disorders) | 1 | 2
Cough (General disorders) | 0 | 1
Body Ache (General disorders) | 0 | 1
Excitement/Agitation (Psychiatric disorders) | 1 | 4
Insomnia (Nervous system disorders) | 1 | 4
Increased Motor Activity (Nervous system disorders) | 0 | 4
Depressive Affect (Psychiatric disorders) | 1 | 2
Headache (Nervous system disorders) | 0 | 2
Drowsiness (Nervous system disorders) | 3 | 1
Decreased Motor Activity (Nervous system disorders) | 2 | 1
Aggression (Psychiatric disorders) | 1 | 1
Akathisia (Nervous system disorders) | 0 | 1
Head Banging (Psychiatric disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Lethargy/Tiredness (Nervous system disorders) | 1 | 0
Nasal Congestion (General disorders) | 4 | 3
Dry Mouth (General disorders) | 3 | 1
Blurred Vision (Eye disorders) | 1 | 1
Ear Infection (Ear and labyrinth disorders) | 1 | 0
Runny Nose (General disorders) | 1 | 0
Sore Throat (General disorders) | 1 | 0
Cold Sore (Skin and subcutaneous tissue disorders) | 1 | 0
Decreased Appetite (Gastrointestinal disorders) | 5 | 4
Nausea/Vomiting (Gastrointestinal disorders) | 2 | 2
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 0
Increased Urination (General disorders) | 1 | 1
Bed Wetting (General disorders) | 0 | 1
Skin Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Bug Bite (Skin and subcutaneous tissue disorders) | 0 | 1
Skin Burn (Skin and subcutaneous tissue disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
The final sample was 83% male and was not statistically powered to detect sex differences in treatment response. Participants were permitted to take other medications during the intervention. Many of our outcome measures relied on parent report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-01-11): https://cdn.clinicaltrials.gov/large-docs/70/NCT01962870/SAP_000.pdf
  • Study Protocol (2016-08-02): https://cdn.clinicaltrials.gov/large-docs/70/NCT01962870/Prot_001.pdf